CLINICAL TRIAL: NCT02075957
Title: Identification by Microarrays of the Risks of Metastatic Relapse, Toxicity and Resistance to Adjuvant Chemotherapy in Completely Resected Non-small Cell Lung Cancer
Acronym: SITRR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2012-A00827-36
Record Dates: First submitted 2014-02-11; First posted 2014-03-03 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer, adjuvant chemo-therapy, DNA chip
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Three blood samples are going to be conserved : one during the week before the operation, one four to eight weeks next to the operation and the last one, at the relapse.
  * Biopsie of non small cell lung cancer will be conserved too.
Oversight: Data Monitoring Committee: No

SUMMARY:
Description of new transcriptional profiles associated with risk of relapse and identification of specific sites of relapse in non-small cell lung cancer, toxicity and resistance to adjuvant chemotherapy in completely resected non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
* A first blood sample will be taken during the week before the operation. A second blood sample will be taken 4 to 8 weeks after the operation. And in case of relapse, a third sample will be taken. These samples are going to be stored in the collection of biological resources of Angers.
* Concerning the biopsy of the resected NSLCL, it will be sent to the collection of biological resources of Angers for conservation directly next to the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Major subject
* Subject who received resection with primary non-small cell lung cancer at the University Hospital of Angers and whose tumor samples will be stored in collection of biological resources of University Hospital of Angers
* A written inform consent.

Exclusion Criteria:

* Under 18 year old;
* Pregnant or nursing women;
* Deprived of liberty;
* Age under curatorship or guardianship;
* Unable to consent person;
* About not carrying a non-small cell lung cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non small cell lung cancer
Sampling Method: Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-01 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Determination of news microarrays profiles of NSCLC relapse risks | 6 to 8 weeks after surgery
  The news microarrays profiles of NSCLC relapse risks will :
  * assessing the risk of relapse in patients undergoing resection of NSCLC (by knowing this risk, patients at highest risk of relapse would be treated as a priority, while avoiding treating patients with low risk)
  * assessing the risk of chemo-resistant tumor cells characters to optimize the choice of treatment to offer to the patient
  * assessing the prediction of sites most likely metastatic relapse to guide survey strategy.
Determination of news microarrays profiles of NSCLC relapse risks | At 1 year
  The news microarrays profiles of NSCLC relapse risks will :
  * assessing the risk of relapse in patients undergoing resection of NSCLC (by knowing this risk, patients at highest risk of relapse would be treated as a priority, while avoiding treating patients with low risk)
  * assessing the risk of chemo-resistant tumor cells characters to optimize the choice of treatment to offer to the patient
  * assessing the prediction of sites most likely metastatic relapse to guide survey strategy.
Determination of news microarrays profiles of NSCLC relapse risks | At 2 years
  The news microarrays profiles of NSCLC relapse risks will :
  * assessing the risk of relapse in patients undergoing resection of NSCLC (by knowing this risk, patients at highest risk of relapse would be treated as a priority, while avoiding treating patients with low risk)
  * assessing the risk of chemo-resistant tumor cells characters to optimize the choice of treatment to offer to the patient
  * assessing the prediction of sites most likely metastatic relapse to guide survey strategy.
Determination of news microarrays profiles of NSCLC relapse risks | At 3 years
  The news microarrays profiles of NSCLC relapse risks will :
  * assessing the risk of relapse in patients undergoing resection of NSCLC (by knowing this risk, patients at highest risk of relapse would be treated as a priority, while avoiding treating patients with low risk)
  * assessing the risk of chemo-resistant tumor cells characters to optimize the choice of treatment to offer to the patient
  * assessing the prediction of sites most likely metastatic relapse to guide survey strategy.
Determination of news microarrays profiles of NSCLC relapse risks | At 4 years
  The news microarrays profiles of NSCLC relapse risks will :
  * assessing the risk of relapse in patients undergoing resection of NSCLC (by knowing this risk, patients at highest risk of relapse would be treated as a priority, while avoiding treating patients with low risk)
  * assessing the risk of chemo-resistant tumor cells characters to optimize the choice of treatment to offer to the patient
  * assessing the prediction of sites most likely metastatic relapse to guide survey strategy.
Determination of news microarrays profiles of NSCLC relapse risks | At 5 years
  The news microarrays profiles of NSCLC relapse risks will :
  * assessing the risk of relapse in patients undergoing resection of NSCLC (by knowing this risk, patients at highest risk of relapse would be treated as a priority, while avoiding treating patients with low risk)
  * assessing the risk of chemo-resistant tumor cells characters to optimize the choice of treatment to offer to the patient
  * assessing the prediction of sites most likely metastatic relapse to guide survey strategy.
Determination of news microarrays profiles of NSCLC relapse risks | At 6 years
  The news microarrays profiles of NSCLC relapse risks will :
  * assessing the risk of relapse in patients undergoing resection of NSCLC (by knowing this risk, patients at highest risk of relapse would be treated as a priority, while avoiding treating patients with low risk)
  * assessing the risk of chemo-resistant tumor cells characters to optimize the choice of treatment to offer to the patient
  * assessing the prediction of sites most likely metastatic relapse to guide survey strategy.
Determination of news microarrays profiles of NSCLC relapse risks | At 7 years
  The news microarrays profiles of NSCLC relapse risks will :
  * assessing the risk of relapse in patients undergoing resection of NSCLC (by knowing this risk, patients at highest risk of relapse would be treated as a priority, while avoiding treating patients with low risk)
  * assessing the risk of chemo-resistant tumor cells characters to optimize the choice of treatment to offer to the patient
  * assessing the prediction of sites most likely metastatic relapse to guide survey strategy.
Determination of news microarrays profiles of NSCLC relapse risks | At 8 years
  The news microarrays profiles of NSCLC relapse risks will :
  * assessing the risk of relapse in patients undergoing resection of NSCLC (by knowing this risk, patients at highest risk of relapse would be treated as a priority, while avoiding treating patients with low risk)
  * assessing the risk of chemo-resistant tumor cells characters to optimize the choice of treatment to offer to the patient
  * assessing the prediction of sites most likely metastatic relapse to guide survey strategy.
Determination of news microarrays profiles of NSCLC relapse risks | At 9 years
  The news microarrays profiles of NSCLC relapse risks will :
  * assessing the risk of relapse in patients undergoing resection of NSCLC (by knowing this risk, patients at highest risk of relapse would be treated as a priority, while avoiding treating patients with low risk)
  * assessing the risk of chemo-resistant tumor cells characters to optimize the choice of treatment to offer to the patient
  * assessing the prediction of sites most likely metastatic relapse to guide survey strategy.
Determination of news microarrays profiles of NSCLC relapse risks | At 10 years
  The news microarrays profiles of NSCLC relapse risks will :
  * assessing the risk of relapse in patients undergoing resection of NSCLC (by knowing this risk, patients at highest risk of relapse would be treated as a priority, while avoiding treating patients with low risk)
  * assessing the risk of chemo-resistant tumor cells characters to optimize the choice of treatment to offer to the patient
  * assessing the prediction of sites most likely metastatic relapse to guide survey strategy.

CONTACTS AND LOCATIONS:
Overall Officials: José HUREAUX, Doctor, Principal Investigator — University Hospital, Angers
Locations (1):
- UH Angers, Angers, Maine et Loire, France